CLINICAL TRIAL: NCT05167188
Title: Prospective Multicenter Study for the Evaluation of GvHD Damage on Medullary Mesenchymal Stem Cells - GvHD Damage on MSCs
Brief Title: Evaluation of GvHD Damage on Medullary Mesenchymal Stem Cells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Prof., Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: GvHD damage on MSCs
Record Dates: First submitted 2021-11-24; First posted 2021-12-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Spontaneous, multicenter, prospective, non-pharmacological study. At the diagnosis of acute or chronic GvHD after HSCT, bone marrow cells will be analysed for MSC content and properties. Bone marrow aspirate will be performed according to usual clinical practise

ELIGIBILITY:
Inclusion Criteria:

* Patients (children and adults) developing acute or chronic GvHD after HSCT.
* Age 6 months- month-99 years,
* Landsky-Karnofsky> 70%,
* Acute or chronic GvHD needing further immunosuppressive treatment.

Exclusion Criteria:

* Anything not included in the inclusion criteria.

Ages: 6 Months to 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients (children and adults) developing acute or chronic GvHD after HSCT
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of damage generated by acute or chronic GvHD on the MSCs after HSCT | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No